CLINICAL TRIAL: NCT00891098
Title: Comparing Imaginal Exposure (IE) and Imagery Rescripting and Reprocessing Therapy (IRRT) in the Treatment of Posttraumatic Stress Disorder (PTSD)
Brief Title: Comparing Imaginal Exposure and Imagery Rescripting in Treatment of Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modum Bad (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Asle Hoffart, phd, Modum Bad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2-Hoffart
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Implosive Therapy; Intermittent Renal Replacement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imaginal exposure (Active Comparator)
  Interventions: Behavioral: Imaginal exposure
- Imagery rescripting (Experimental)
  Interventions: Behavioral: Imagery rescripting

INTERVENTIONS:
Behavioral: Imaginal exposure — 7 individual sessions of imaginal exposure of trauma memories according to the prolonged exposure treatment manual
  Other Names: prolonged exposure; pe
  Arms: Imaginal exposure
Behavioral: Imagery rescripting — 7 individual sessions of imagery rescripting of trauma memories according to the imagery rescripting and reprocessing therapy manual
  Other Names: rescripting; irrt
  Arms: Imagery rescripting

SUMMARY:
The outcome of trauma treatment (Posttraumatic Stress Disorder - PTSD) may be influenced by which emotions that are predominant among current symptoms, e.g. fear, anger, guilt, shame. Different treatment procedures for processing traumatic memories may resolve different emotions. This study compares two different treatment procedures of working with trauma memories in PTSD treatment (namely, Imaginal Exposure and Imagery Rescripting) in order to test this.

DETAILED DESCRIPTION:
The main objectives of this study are:

1. To assess the relative efficacy of the two procedures in inpatient treatment for PTSD
2. To assess whether the predominant emotions in the traumatic memories moderate the outcome of the different procedures
3. To assess whether theory-derived constructs mediate outcome and whether the mediating relationships are different in the two treatments
4. To provide a theoretical account of the two models
5. To psychometrically evaluate 3 new measures

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of PTSD identified as primary diagnosis
* Accepts withdrawal of all psychotropic medication

Exclusion Criteria:

* Extensive dissociative symptoms or current psychosis,
* Current suicidal risk,
* Extensive current substance or alcohol abuse, or
* Ongoing trauma

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms | pretreatment, weekly during treatment, posttreatment, followup

SECONDARY OUTCOMES:
General psychiatric symptoms | pretreatment, weekly during treatment, postttreatment, followup

CONTACTS AND LOCATIONS:
Overall Officials: Asle Hoffart, PhD, Study Chair — Modum Bad and University of Oslo
Locations (1):
- Modum Bad, Vikersund, Buskerud, Norway